CLINICAL TRIAL: NCT06719648
Title: Multiple Gingival Recessions Root Coverage Using Coronally Advanced Tunnel Technique Combined with a Xenogenic Dermal Matrix (Novomatrix®): a Randomized Clinical Trial
Brief Title: Root Coverage for Gingival Recessions: a Randomized Clinical Trial Using Coronally Advanced Tunnel Technique and Novomatrix®
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Andres Pascual La Rocca, Periodontist, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PER-ECL-2019-07; PER-ECL-2019-07 (Other: Universidad Internacional de Catalunya)
Record Dates: First submitted 2024-11-14; First posted 2024-12-06 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: L-PRF; Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Novomatrix and LPRF (Experimental): Incisions: Incisions were made in the gums using a specialized scalpel. Flap Elevation: The gum tissue was lifted away from the underlying bone using a dental elevator.
  Partial Thickness Dissection: The tissue was cut to release tension and allow for easier repositioning.
  Interdental Papilla Elevation: The gum tissue between the teeth was partially lifted.
  Flap Extension: The flap was extended to cover more teeth for better coverage. Tissue Separation: The flap was carefully separated from underlying tissues to allow for proper positioning.
  Root Preparation: The exposed root surfaces were smoothed and cleaned.
  Interventions: Device: Acellular dermal matrix + L-Prf
- Connective tissue graft and LPRF (Active Comparator): Incisions: Incisions were made in the gums using a specialized scalpel. Flap Elevation: The gum tissue was lifted away from the underlying bone using a dental elevator.
  Partial Thickness Dissection: The tissue was cut to release tension and allow for easier repositioning.
  Interdental Papilla Elevation: The gum tissue between the teeth was partially lifted.
  Flap Extension: The flap was extended to cover more teeth for better coverage. Tissue Separation: The flap was carefully separated from underlying tissues to allow for proper positioning.
  Root Preparation: The exposed root surfaces were smoothed and cleaned.
  Interventions: Procedure: Connective Tissue graft + L-Prf

INTERVENTIONS:
Device: Acellular dermal matrix + L-Prf — Incisions: Incisions were made in the gums using a specialized scalpel. Flap Elevation: The gum tissue was lifted away from the underlying bone using a dental elevator.
  Partial Thickness Dissection: The tissue was cut to release tension and allow for easier repositioning.
  Interdental Papilla Elevation: The gum tissue between the teeth was partially lifted.
  Flap Extension: The flap was extended to cover more teeth for better coverage. Tissue Separation: The flap was carefully separated from underlying tissues to allow for proper positioning.
  Root Preparation: The exposed root surfaces were smoothed and cleaned.
  Arms: Novomatrix and LPRF
Procedure: Connective Tissue graft + L-Prf — Incisions: Incisions were made in the gums using a specialized scalpel. Flap Elevation: The gum tissue was lifted away from the underlying bone using a dental elevator.
  Partial Thickness Dissection: The tissue was cut to release tension and allow for easier repositioning.
  Interdental Papilla Elevation: The gum tissue between the teeth was partially lifted.
  Flap Extension: The flap was extended to cover more teeth for better coverage. Tissue Separation: The flap was carefully separated from underlying tissues to allow for proper positioning.
  Root Preparation: The exposed root surfaces were smoothed and cleaned.
  Arms: Connective tissue graft and LPRF

SUMMARY:
A randomized clinical trial comparing the modified tunnel technique with the use of acellular xenogeneic matrix and connective tissue with the use leucocyte platlet rich fibrin (L-PRF)

DETAILED DESCRIPTION:
Study design In the pre-surgical clinical evaluation periodontal measurements were registered at baseline and during the follow-up period: periodontal probing depth (PPD), clinical attachment level (CAL), width and length (mm) of the GR, type of GR, amount of attached gingiva (mm), depth of vestibule (mm), interdental papilla height (mm), non carious cervical lesions, visual LAC detection, gingival thickness (mm) and gingival phenotype (translucency of the periodontal probe). Intraoral photographs always showing a frontal view of the treated area were taken. Moreover, all patients received supragingival scaling and crown polishing. Patient were instructed to rinse with 0.12% Chlorhexidine, 2 times a day for 1 minute starting one week prior to the surgery. Local etiological factors in the area of treatment were controlled or modified, such as the removal and change of overflowing seals, the polishing of restorations, the adjustment of margins. In cases where the cement enamel junction is not clearly detected a reconstruction of this with resin was carried out. Finally, prior to surgery, anti-inflammatory treatment were prescribed to the patient from the day before surgery with Ibuprofen 400 mg, 1 every 8 hours for 7 days

Clinical Procedures:

Prior to surgical procedure, a sealed envelope was opened with the treatment modality (randomization table). Local infiltration anesthesia was performed on both sides (buccal and lingual/palatal) of the affected area. The surgical protocol was performed following the tunnel technique described by Allen (1994) and using microsurgical instruments for periodontal plastic surgery [KPA Allen, PPAELA, tunelisation knife black line, (Hu Fredy)]. The flap was exposed using a modified coronal tunnel technique with partia papillae elevation.

The protocol was started with intra-muscular incisions with an intrasurcular scalpel (KPA Allen) in each of the treated teeth. Elevation of the flap was performed, using the Allen elevator (PPAELA), till the mucogingival line. After reaching this limit, a partial thickness dissection started using the modified Orban knife, until full tension of the flap was eliminated. The interdental papilla's was partially elevated, without being cut from their alveolar base in order to be able to coronally advance the flap to a coronal position free from tension. The flap was extended one tooth mesial and one tooth distal of the treatment area. The separation of the flap from small muscle fibers and bundles of collagen fibers was carefully carried out until the flap can passively be positioned at least 1mm above the cement enamel junction of all the involved teeth, in order to ensure the passive reposition of the flap and the posterior suture free of tension. After assuring the adequate extension of the tunnel, preparation and decontamination of the roots was carried out using Gracey curettes, eliminating the superficial cement surface in relation to the exposed root portion in order to achieve a smooth and flat surface.

All clinical procedures were performed by the same experienced surgeon who was blind to the treatment modality. All evaluations, procedures and controls will be performed in the dental center and pavilions of the Clinic of the Universidad de los Andes and the International University of Cataluña, were two experienced peridontontis (A.C and A.P) will perform the MCAT.

L-PRF procedure protocol Before the beginning of the surgery, 4 tubes of blood without anticoagulant were taken to obtain the L-PRF. This tubes were filled by venous puncture with a butterfly of diameter 24, they were immediately centrifuged at a speed of 2700 rpm for a period of 12 minutes. The tubes were removed from the centrifuge and the result is a fibrin clot with a platelet content located between a layer of lower red blood cells and acellular plasma on the surface, this clot was removed from the tube and the red blood cells adhering to it are removed and discarded. In continuation, the L-PRF clot was placed in a PRF Box (Process Ltd., Nice, France), where it is covered with a compressor. After approximately 1 minute the result is a membrane or autogenous fibrin matrix. Both the Novomatrix matrix and the connective graft will be left in a cup with part of the plasma exudate resulting from the manufacture of the fibrin matrix for a couple of minutes and will be injected with this biological product by injection with tuberculin syringe once positioned under the tunneled flap.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Presence of 2 or more adjacent Cairo's type I or II gingival recessions
* Non-smokers
* Plaque index <20% and bleeding on probing (BOP) <20%
* Periodontal health
* Existing endodontic therapies must be carefully evaluated. In case of inadequate treatments, endodontic retreatment will be performed (i.e., a minimum of two months before performing the surgical therapy).
* Use of optical magnification (2.5X) and microsurgical instruments for the surgical procedure is recommended.

Exclusion Criteria:

* Individuals who do not meet the inclusion criteria
* Systemic compromise involving healing response and tissue repair, or coagulation disorders
* Uncontrolled systemic diseases
* Use of anticoagulant therapy or bisphosphonates
* Active periodontal disease
* Inadequate psychological profile
* Patients with intentions to change residence that would prevent follow-up
* Multiple recessions in molars

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2020-05-20 (Actual); Primary Completion 2023-04-27 (Actual); Study Completion 2024-04-28 (Actual)

PRIMARY OUTCOMES:
Mean root coverage | Baseline, 6 and 12 months
  amount of root surface covered by healthy gum tissue

SECONDARY OUTCOMES:
Complete root coverage | Baseline, 6 and 12 months
  all of the exposed root surface of a tooth has been fully covered by healthy gum tissue

CONTACTS AND LOCATIONS:
Locations (1):
- Isabel Arroyo, Barcelona, Barcelona, Spain